CLINICAL TRIAL: NCT05209009
Title: A Randomized, Observer-Blind, Dose-Escalation Phase 2 Clinical Trial of COVAC-2 in Generally Healthy Adults
Brief Title: A Clinical Trial of COVAC-2 in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Government of Canada (Other Government); Government of Saskatchewan (Other Government); Vaccine Formulation Institute (VFI) (Unknown); Seppic (Industry)
Responsible Party: Principal Investigator, Volker Gerdts, Director & CEO, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COVAC-003
Record Dates: First submitted 2021-12-02; First posted 2022-01-26 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2
MeSH Terms: interventions — COVAC-1 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): COVAC-2 25 µg: 200 generally healthy adults > 18 years of age receive the vaccine on Day 0, followed by a second dose on Day 28.
  Interventions: Biological: COVAC-2
- Group B (Placebo Comparator): 100 generally healthy adults > 18 years of age receive a dose of normal saline (placebo) on Day 0, followed by a dose of normal saline (placebo) on Day 28.
  Interventions: Biological: Saline Placebo

INTERVENTIONS:
Biological: COVAC-2 — Intramuscular vaccine against SARS-CoV-2
  Arms: Group A
Biological: Saline Placebo — Intramuscular injection of saline placebo
  Arms: Group B

SUMMARY:
VIDO has developed a vaccine called COVAC-2.

The COVAC-2 study vaccine contains a portion of the SARS-CoV-2 spike protein, called S1. The spike protein is the part of the virus that is responsible for attaching to the surface of host cells. COVAC-2 contains a SWE adjuvant. An adjuvant is a compound that is added to a vaccine to help the vaccine produce a better immune response. The SWE adjuvant is similar to another adjuvant, MF59, that is found in influenza vaccines and MF59 containing vaccines have been given to millions of people around the world. The vaccine is expected to stimulate the body to make antibodies against the S1 protein. The antibodies will recognize the viral spike protein if the body is exposed to the virus and prevent severe COVID-19 illness. In animal studies, the immune response generated by the COVAC-2 vaccine was able to protect the vaccinated animals against a severe SARS-CoV-2 infection.

This is a Phase 2, placebo-controlled, observer-blind, age-stratified randomized, multicentre study to test the safety and immunogenicity of a dose level of the COVAC-2 vaccine (25 µg protein) administered twice (4 weeks apart) in generally healthy adults 18+ years of age. Up to 300 participants will be enrolled. For an individual participant, the duration of study will be approximately 12 months from the first vaccination (Day 0).

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy male and female adults aged 18 years of age or older at the time of signing the informed consent form;
2. Good general health as determined by screening evaluation not greater than 30 days before injection of first dose;

   Note: Participants who are overtly healthy as determined by medical evaluation or are considered medically stable according to the judgment of the investigator. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalisation for worsening disease during the 3 months prior to enrolment, and/or hospitalization within the entire study period is not anticipated. Also, the participant appears likely to be able to remain in follow-up through the end of protocol-specified period. Mild to moderate well-controlled comorbidities are allowed.
3. If female of child-bearing potential and heterosexually active, practice of adequate contraception for 30 days prior to injection, negative pregnancy test on the day of injection, and agreement to continue adequate contraception until 180 days after the second injection;
4. Male participants are eligible to participate in the study if they agree to the following requirements during the study period and for at least 28 days after the last injection of study dose, i.e.,

   o Be abstinent from any heterosexual intercourse with a female of childbearing potential as their preferred and usual lifestyle.

   OR

   o Must agree to use a male condom when engaging in any activity that allows for passage of ejaculate to another person. In addition to male condom use, a highly effective method of contraception should be considered in women of child-bearing potential partners of male participants.

   AND

   o Must refrain from donating sperm; and
5. Written informed consent, after review of the consent form and having adequate opportunity to discuss the study with an investigator or a qualified designee and pass the "Test of Understanding" (up to 3 attempts). For participants who cannot read or write, the consent must be witnessed by a literate third party not involved in study conduct.

Exclusion Criteria:

1. Presence of any febrile illness or any known or suspected acute illness on the day of any immunization;
2. Clinically significant bleeding disorder (e.g., clotting factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture.
3. Any condition, which in the opinion of the Investigator, may make the participant inappropriate for the study;
4. Receiving systemic immunosuppressive therapy or history of receiving chemotherapy in last 5 years other than topical agents;
5. Receipt of systemic glucocorticoids (a dose ≥ 20 mg/day prednisone or equivalent for 14 days) within 1 month, or any other cytotoxic or immunosuppressive drug within 6 months;
6. Cancer diagnosis in the last 5 years, excluding basal cell and squamous cell carcinoma of the skin, which are allowed;
7. Presence of autoimmune disease;
8. Receipt of any investigational drug within 6 months;
9. Receipt of any non-COVID-19 authorized vaccines within 2 weeks of receiving study dose injection;
10. Receipt of any authorized COVID-19 vaccine prior to study enrollment;
11. Receipt of any other experimental SARS-CoV-2/COVID-19 or other experimental coronavirus vaccine(s) at any time prior to or during the study;
12. Receipt of blood products or immunoglobulin (IVIg or IMIg) within 3 months of study entry/baseline serologic evaluation;
13. Current anti-tuberculosis therapy;
14. History of any reaction or hypersensitivity likely to be exacerbated by any component of the study vaccine;
15. Hematologic or biochemical laboratory abnormalities (blood or urine), as defined by lab normal ranges. To exclude transient abnormalities, the investigator may repeat a test once, and if the repeat test is normal according to local reference ranges, participant may be enrolled. Grade 1 abnormalities of laboratory values will not be exclusionary if considered not clinically significant by the investigator; and
16. Pregnant and breastfeeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the safety and tolerability of COVID-19 vaccine (COVAC-2) following two consecutive injections (28 days apart) in generally healthy volunteers | Up to 365 days
  Incidence of solicited adverse events (AE) up to 7 days post-injection; unsolicited AEs up to 28 days post-injection; any clinically significant laboratory up to 28 days post-injection; and any serious AEs (SAEs), medically attended events (MAE), or Adverse Event of Special Interest (AESI) up to Day 365.

SECONDARY OUTCOMES:
To assess the induction of SARS-CoV-2 spike protein (S) antibodies following two consecutive injections (28 days apart) of COVAC-2 vaccine through use of Enzyme-Linked immunosorbent Assay (ELISA) up to Day 365 | Up to 365 days
  SARS-CoV-2 specific antibodies to Wuhan spike antigen or pseudovirus neutralizing antibodies pre- injection and post-injection as measured by spike protein-specific ELISA and serum neutralization assay.
To assess SARS-CoV-2 spike protein-specific, cell-mediated response up to Day 365 induced by two consecutive injections (28 days apart) of COVAC-2 vaccine | Up to 365 days
  Measurement of SARS-CoV-2 spike protein-specific, cell-mediated response markers in Peripheral Blood Mononuclear Cells (PBMCs) pre- and post-injection.

OTHER OUTCOMES:
To evaluate the level of neutralizing antibody response against SARS-CoV-2 variants of concern (VOCs) up to Day 365 induced by two consecutive injections (28 days apart) of COVAC-2 vaccine | Up to 365 days
  Neutralizing antibodies against SARS-CoV-2 VOCs pre- injection and post-injection as measured by serum neutralization assay.

CONTACTS AND LOCATIONS:
Locations (2):
- Uganda (2):
  - Uganda Virus Research Institute, Entebbe
  - Epicentre, Mbarara Research Centre, Mbarara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garg R, Liu Q, Van Kessel J, Asavajaru A, Uhlemann EM, Joessel M, Hamonic G, Khatooni Z, Kroeker A, Lew J, Scruten E, Pennington P, Deck W, Prysliak T, Nickol M, Apel F, Courant T, Kelvin AA, Van Kessel A, Collin N, Gerdts V, Koster W, Falzarano D, Racine T, Banerjee A. Efficacy of a stable broadly protective subunit vaccine platform against SARS-CoV-2 variants of concern. Vaccine. 2024 Aug 13;42(20):125980. doi: 10.1016/j.vaccine.2024.05.028. Epub 2024 May 19. PMID 38769033